CLINICAL TRIAL: NCT01873885
Title: Phase 1, Randomized, Double-Blind, Placebo-Controlled Exploratory Study That Will Assess the Safety, Tolerability, Pharmacokinetics and Hemodynamic Response to a Single 30 Minute Intravenous Infusion of Vasomera™ (PB1046) in Adult Subjects With Stage 1 or 2 Essential Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PhaseBio Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: PB1046-PT-CL-0002
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Essential Hypertension
Keywords: PB1046, VIP, Essential Hypertension, Vasomera
MeSH Terms: conditions — Essential Hypertension | interventions — VIP-ELP fusion molecule PB1046

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1: Single IV Infusion Vasomera (PB1046) or Placebo (Experimental): Cohort 1 - Single 30 minute infusion Vasomera (PB1046) at 0.01 mg/kg diluted in 0.9% Sodium Chloride or Placebo (0.9% Sodium Chloride)
  Interventions: Drug: Placebo Single IV (Intravenous) Infusion; Drug: Experimental: Single IV Infusion Vasomera (PB1046)
- Cohort 2: Single IV Infusion Vasomera (PB1046) or Placebo (Experimental): Cohort 2 - Single 30 minute infusion Vasomera (PB1046) at 0.005mg/kg in 0.9% Sodium Chloride or Placebo (0.9% Sodium Chloride)
  Interventions: Drug: Placebo Single IV (Intravenous) Infusion; Drug: Experimental: Single IV Infusion Vasomera (PB1046)
- Cohort 3: Single IV Infusion Vasomera (PB1046) or Placebo (Experimental): Cohort 3 - Single 30 minute infusion Vasomera (PB1046) at 0.02mg/kg 0.9% Sodium Chloride or Placebo (0.9% Sodium Chloride)
  Interventions: Drug: Placebo Single IV (Intravenous) Infusion; Drug: Experimental: Single IV Infusion Vasomera (PB1046)

INTERVENTIONS:
Drug: Placebo Single IV (Intravenous) Infusion — 0.9% Sodium Chloride - 30 minute IV infusion
Drug: Experimental: Single IV Infusion Vasomera (PB1046)

SUMMARY:
This study is an exploratory Phase 1 randomized, double-blind (Investigator and study subject and 2-D echo endpoint assessor), placebo-controlled single IV infusion dose escalation study that will enroll up to approximately 32 subjects with stage 1 or 2 essential hypertension.

DETAILED DESCRIPTION:
The study will be conducted in two parts.

Part 1: For the initial evaluation of safety, pharmacokinetic exposure and pharmacodynamic response, subjects will be tapered off antihypertensive background therapy.The initial starting dose will be a sub-therapeutic dose. Dose escalation will continue with a maximum of a doubling of the previous dose until either 1) a maximum tolerated dose (MTD) is identified or 2) modeling of the pharmacokinetic (PK) data indicate that maximum exposure (Cmax) at the next planned dose level would exceed a maximum drug concentration (Cmax) which was the maximum observed drug concentration following a single subcutaneous administration in Study PB1046-PT-CL-0001.

Part 2: The dose group which is capable of providing a Cmax exposure which is capable of eliciting a clinically relevant hemodynamic response, will be expanded to enroll an additional 12 subjects (6 active and 6 placebo).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign a written informed consent and follow all study related procedures.
* Males or females age 18 - 80 years of age inclusive.
* Male and female subjects of childbearing potential must be willing and able to practice effective contraception during the study, and be willing and able to continue contraception for 1 month (30 days) after their last dose of study drug.
* BMI ≥ 20 but ≤ 40 kg/m2
* Diagnosed with essential hypertension and are currently taking one or more antihypertensive medications to control their blood pressure and, who in the opinion of the investigator, could be safely withdrawn from antihypertensive therapy.

Exclusion Criteria:

* Known allergy to the study drug or any of its components, or who have previously received Vasomera (PB1046).
* Inadequate "imaging window" by echocardiography as determined by screening echocardiography (core assessment), or cardiac abnormalities that may confound echocardiography readings (i.e., mitral regurgitation, "floppy-valve" syndrome) for evaluation of secondary study endpoints.
* Seated systolic blood pressure <120 mmHg or diastolic blood pressure < 80 mmHg (confirmed in triplicate) at randomization (Day -1) or prior to the first dose of study drug (V3 Day 0) will exclude the subject from participation.
* Evidence of sustained elevation in systolic blood pressure >169 mmHg or diastolic blood pressure >109 mmHg prior to dosing (Day 0) during the washout period which in the opinion of the investigator would place the subject at risk for continued study participation (i.e., can not be safely withdrawn from antihypertensive therapy).
* Clinically significant changes in health status or concomitant prescription medications within 2 weeks prior to dosing (V3 Day 0) that could place the subject at risk for dosing with study drug or confound the primary or secondary outcome measures as assessed by the Investigator.
* Unstable/underlying cardiovascular disease defined as: a. Congestive heart failure (NYHA class III-IV), stroke, transient ischemic attack, unstable angina pectoris, or myocardial infarction within the 6 months prior to screening (V1) b. Mean triplicate 12-lead ECG demonstrating a QT interval (corrected using Fridericia's formula (QTcF)) >450 msec in males and >470 msec in females at Screening, (V1) or a history or evidence of long QT syndrome. c. Sustained heart rate >100 beats per minute (BPM) (at rest) at screening (V1), prior to randomization (V3 Day -1), or prior to dosing (V3 Day 0). d. Any episode of atrial fibrillation, ventricular tachycardia (defined as ten (10) or more beats with heart rate greater than 130 beats per minute), ventricular fibrillation, firing of an implantable cardiac defibrillator (ICD) for documented ventricular ectopy, or other clinically significant documented arrhythmias within 3 months prior to administration of study drug (V3 Day 0).
* Uncontrolled diabetes defined as a Hemoglobin A1c > 10.0%. Note: only applicable for subjects with a known or suspected history of diabetes.
* Clinically significant renal and/or hepatic dysfunction at Screening (V1) or at baseline (V3 Day -1).
* Pregnant or lactating females.
* Known history of or active drug or alcohol abuse within the 12 months prior to screening (V1) and/or positive drug screen (for illicit drugs) or detection of alcohol at baseline.
* Positive for Human Immunodeficiency Virus (HIV) antibodies, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies.
* Participation in any other study and have received any other investigational drug or device within 30 days prior to the Screening visit or are taking part in a non-drug study which in the opinion of the Investigator would interfere with the outcome of the study.
* Major surgery, donated or lost > or = 1 unit of blood (approximately 500 mL) within 30 days prior to Screening (V1) or display evidence of volume depletion (i.e., postural hypotension) prior to randomization (V3 Day -1) or dosing (V3 Day 0).
* Other medical or psychiatric condition which in the opinion of the Investigator would place the subject at increased risk, would preclude obtaining voluntary consent, or would confound the results of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Days -45 to 28: Vital signs (Days -45, -14, -1, 0, 1, 2, 3, 4, 7, 14 and 28), ECGs (Days -45, -1, 0, 1 and 2), Safety Labs (Days -45, -1, 1, 7 and 28), and Telemetry (Days -1, 0 and 1)
  To evaluate the safety and tolerability of single ascending doses of Vasomera administered as a 30 minute intravenous (IV) infusion to subjects with stage 1 or stage 2 essential hypertension.
  * Incidence and severity of adverse events (AEs) and their relationship to Vasomera (including AEs of interest, i.e., incidence and severity of gastrointestinal effects, and infusion site reactions)
  * Changes in vital signs, ECGs, safety laboratory parameters, heart rhythm via telemetry monitor from baseline
Pharmacokinetic Profile | Days 0, 1, 2, 3, and 4
  To evaluate the pharmacokinetic profile of single ascending doses of Vasomera administered as a 30 minute intravenous (IV) infusion to subjects with stage 1 or stage 2 essential hypertension.
  * Elimination Half-life (t½)
  * Area under the concentration curve from time 0 to infinity (AUC0-inf)
  * Area under the curve to the final sample
  * Time to maximum concentration (Tmax)
  * Maximum serum concentration (Cmax)
  * Elimination rate constant (Lambda-z)
  * Clearance (CL)
  * Distribution (Vz)
  * Compartmental modeling - If the graphical presentations of the individual subject serum concentrations vs. time suggest that a compartmental model may be consistent with the data, then an appropriate compartmental model will be fit to the data.

SECONDARY OUTCOMES:
Hemodynamic Parameters | Days -14, 0, 1, 2, 3, 4, 7, 14 and 28
  Compare changes in hemodynamic parameters as measured by serial systolic and diastolic blood pressure (BP) measurements and echocardiography compared to placebo.
  Change from baseline in systolic and diastolic BP and heart rate (HR).
  Change from baseline in two-dimensional echocardiography parameters which may include:
  * BP and HR
  * Left ventricular (LV) internal diameter in diastole and in systole, wall thickness in diastole, outflow tract diameter in mid-systole, volumes in end-diastole and end-systole, and outflow tract flow-time velocity integral
  * Ascending aorta peak flow velocity
  * Transmitral flow velocity pattern
  * Doppler tissue imaging of tricuspid, septal and mitral annulus
  * Left atrial volume
  * Derivation of: LV Ejection Fraction, LV Stroke Volume and Index, LV Cardiac Output and Index, Ejection Time, Systemic Vascular Resistance, Mitral E and A velocities, LV and index, Myocardial tissue velocities S' and e'.
Immunogenicity Assessment | Days 0, 14 and 28
  Evaluate if subjects elicit an immune response to study drug and if that response cross reacts with related endogenous compounds following a single 30 minute IV infusion.

CONTACTS AND LOCATIONS:
Overall Officials: William B. Smith, MD, Principal Investigator — New Orleans Center for Clinical Research- Knoxville
Locations (1):
- New Orleans Center for Clinical Research - Knoxville, Knoxville, Tennessee, United States